CLINICAL TRIAL: NCT04990089
Title: VIVO in a Practical Clinical Experience
Brief Title: VIVO European Observational Registry
Status: Completed | Type: Observational
Sponsor: Catheter Precision. Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 02-0521-001
Record Dates: First submitted 2021-07-27; First posted 2021-08-04 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Ventricular Arrythmia; Ventricular Tachycardia; Premature Ventricular Contraction
MeSH Terms: conditions — Tachycardia, Ventricular; Ventricular Premature Complexes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: VIVO — VIVO is a per-procedural planning tool designed to non-invasively identify the origin of a ventricular arrhythmia.

SUMMARY:
A multi-center, observational registry conducted in Europe and the UK to prospectively review VIVO in a clinical setting in 125 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients must at least 18 years of age Patients who have signed an IRB/EC approved patient informed consent and applicable patient privacy protection authorization per local law
* Patients who have previously had contrast cardiac imaging or will have cardiac imaging ordered per standard of care
* Patients will be selected without regard to gender.

Exclusion Criteria:

• Patients that are unable to receive contrast cardiac imaging (MR or CT)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients experiencing ventricular tachycardia (VT) or premature ventricular contractions (PVC) and being considered for or have a scheduled a ventricular ablation procedure.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2021-10-21 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-09-28 (Actual)

PRIMARY OUTCOMES:
Measure the effectiveness of VIVO within different types of VA procedures | 1 day
  The primary effectiveness objective is to assess the types of procedures where VIVO is used to plan and/or guide the ablation procedure or to determine a diagnosis of arrhythmia.
  Primary Effectiveness endpoint: Summarize the types of procedures where VIVO was utilized in the procedure to include the number of VT vs PVC, whether VIVO improved procedural planning and acute procedural success measured as termination or reduction in arrhythmia.
Measure the safety by observing adverse events related to the device and procedure | 1 day
  Primary safety objective is to assess any adverse events related to the device and procedure.
  Primary Safety endpoint: Summarize the number of adverse events related to VIVO or procedure.

SECONDARY OUTCOMES:
Effectiveness | 12 months
  Secondary effectiveness objective is to evaluate the success of the ablation procedure (if performed) at follow- up visits (3, 6 and 12 months).
  Secondary effectiveness endpoint: Summarize the success of the ablation procedure at each follow up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Andre Ng, MD, Principal Investigator — Glenfield University Hospital
Locations (8):
- Mater Private Hospital, Dublin, Ireland
- Mazzoni Hospital, Ascoli Piceno, Italy
- Netherlands (2):
  - University Medical Center Groningen, Groningen
  - Erasmus Medical Center, Rotterdam
- La Luz Hospital, Lisbon, Portugal
- United Kingdom (3):
  - Glenfield University Hospital, Leicester
  - Royal Brompton Hospital, London
  - John Radcliffe University Hospital, Oxford

IPD SHARING:
Plan to Share IPD: No
NO IPD is to be shared with other researchers.